CLINICAL TRIAL: NCT06588400
Title: AOSEPT™ PLUS With HydraGlyde FID 120947A and AOCup Lens Case (CLEAR CARE PLUS) and AOSEPT™ PLUS FID 119056 and AOCup Lens Case (CLEAR CARE) Family PMCF Study
Brief Title: AOSEPT (CLEAR CARE) PLUS Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LCT783-P001
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Contact Lens Care
Keywords: Contact Lens Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- AOSEPT Plus (CC) (Experimental): AOSEPT Plus and AOCup lens case used as instructed with habitual contact lenses for 90 days. It is expected that the habitual contact lenses will be worn for at least 8 hours per day for at least 5 days per week during study participation.
  Interventions: Device: AOSEPT Plus and AOCup lens case; Device: Habitual contact lenses
- AOSEPT Plus with HydraGlyde (CCP) (Experimental): AOSEPT Plus with HydraGlyde and AOCup lens case used as instructed with habitual contact lenses for 90 days. It is expected that the habitual contact lenses will be worn for at least 8 hours per day for at least 5 days per week during study participation.
  Interventions: Device: AOSEPT Plus with HydraGlyde and AOCup lens case; Device: Habitual contact lenses

INTERVENTIONS:
Device: AOSEPT Plus and AOCup lens case — Commercially available cleaning, disinfecting, and storage system consisting of a hydrogen-peroxide based solution (AOSEPT Plus) and a lens case (AOCup) with a neutralizer disc. The solution and lens case must be used together.
  Other Names: Clear Care (CC)
  Arms: AOSEPT Plus (CC)
Device: AOSEPT Plus with HydraGlyde and AOCup lens case — Commercially available cleaning, disinfecting, and storage system consisting of a hydrogen-peroxide based solution (AOSEPT Plus with HydraGlyde) and a lens case (AOCup) with a neutralizer disc. The solution and lens case must be used together.
  Other Names: Clear Care Plus (CCP)
  Arms: AOSEPT Plus with HydraGlyde (CCP)
Device: Habitual contact lenses — Daily wear, reusable, soft (including hydrogel and silicone hydrogel) or rigid gas permeable (RGP) contact lenses according to subject's habitual prescription worn in both eyes and removed prior to sleep for cleaning and disinfection with the study product provided.

SUMMARY:
The purpose of this post-market clinical follow-up (PMCF) study is to evaluate the long-term safety and performance of 2 commercially available contact lens cleaning and disinfecting systems in a pediatric population.

DETAILED DESCRIPTION:
Subjects will participate in the study for approximately 90 days, with telephone calls scheduled on Day 30 ± 7 (Visit 2) and Day 60 ± 7 (Visit 3) and an in-office follow-up visit scheduled on Day 90 ± 7 (Visit 4). Subjects may have unscheduled visits if deemed necessary per the Investigator's judgment.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject and parent/legally authorized representative able to understand and sign an Institution Review Board approved informed consent/assent form.
* Subject willing to follow and be able to attend all scheduled study visits as required per protocol.
* Successful wear of daily wear, reusable, soft (including hydrogel and silicone hydrogel) or rigid gas permeable (RGP) contact lenses in both eyes for the past 3 months for a minimum of 5 days per week and 8 hours per day.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any ocular disease or condition that would contraindicate contact lens wear.
* Use of systemic or ocular medication that would contraindicate contact lens wear.
* Any known sensitivity to any ingredients in the study products.
* Current or history of pathological dry eye in either eye that would in the opinion of the Investigator preclude contact lens wear.
* Any use of habitual/prescribed topical ocular medication or artificial tear or rewetting drop (habitual) that would require instillation during the study.
* Other protocol-specified exclusion criteria may apply.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Front surface deposits at Day 90 | Day 90
  Protein and lipid deposits on the front surface of the contact lens will be assessed by the investigator using a biomicroscope, which magnifies the appearance of the contact lens on the wearer's eye. Deposits will be graded on a 5-point scale, with 0 being absent and 4 being severe.
Back surface deposits at Day 90 | Day 90
  Protein and lipid deposits on the back surface of the contact lens will be assessed by the investigator using a biomicroscope, which magnifies the appearance of the contact lens on the wearer's eye. Deposits will be graded on a 5-point scale, with 0 being absent and 4 being severe.
Incidence of corneal infiltrative events | Up to Day 90
  A corneal infiltrate is a single or group of inflammatory cells in the normally clear cornea. Corneal infiltrative events will be detected by the investigator during an eye exam.
Incidence of microbial keratitis | Up to Day 90
  Microbial keratitis is a sight-threatening infection of the cornea. Incidences of microbial keratitis will be detected by the investigator during an eye exam.
Incidence of solution induced corneal staining (SICS) | Up to Day 90
  Corneal staining determined by the investigator to be solution-related will be graded by type (pattern of staining) and area (how much) in each of the 5 corneal regions: central, superior, nasal, inferior, temporal.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No